CLINICAL TRIAL: NCT05653713
Title: A Phase 1b, Randomized, Double-blind, Placebo-controlled Study in Healthy Volunteers to Investigate the Effects of CSL324 in the Lung After Segmental Challenge With Endotoxin
Brief Title: Effects of CSL324 in the Lung After Segmental Challenge
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CSL324_1004; 2022-002404-20 (EudraCT Number)
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSL324 (Experimental): Intravenous (IV) dose of CSL324
  Interventions: Drug: CSL324
- Placebo (Placebo Comparator): IV dose of 0.9% saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CSL324 — Single intravenous (IV) dose of CSL324
  Other Names: Recombinant anti-granulocyte colony-stimulating factor (G-CSF) receptor monoclonal antibody (mAb)
  Arms: CSL324
Drug: Placebo — IV dose of 0.9% saline
  Arms: Placebo

SUMMARY:
This is a phase 1b, randomized, double-blind, placebo-controlled study in healthy volunteers to investigate the antiinflammatory effect of pretreatment with CSL324 on response to a lipopolysaccharide (LPS) endotoxin challenge in a single lung segment. Saline will be instilled into a segment in the contralateral lung for the purpose of comparison.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteer.
* Between the ages of ≥ 18 and ≤ 65 years.
* Body mass index within the range of 18 to 32 kg/m2
* Female of nonchildbearing potential or of childbearing potential and willing to use a highly effective method of contraception (in addition to male partner condom with or without spermicide)
* Nonsmoker or an ex-smoker who has stopped smoking (including e-cigarettes or vaping devices) for > 1 year with a smoking history of < 10 pack-years.

Exclusion Criteria:

* Any clinically significant abnormalities in physical examination findings, electrocardiogram (ECG) readings, safety laboratory test results, or ANC < 2.0 × 109 cells/L.
* History of myeloproliferative or lymphoproliferative disease.
* Current or previous history of any immunosuppressive condition.
* Currently receiving any immunosuppressive or immunomodulatory therapy, or history of undergoing such therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Percent reduction in mean absolute neutrophil cell counts in bronchoalveolar lavage fluid (BALF) between CSL324 and placebo | Obtained at 24 hours after the segmental lipopolysaccharide (LPS) challenge with endotoxin in the lung

SECONDARY OUTCOMES:
Percent reduction in the mean change in biomarkers of neutrophil activation in BALF from Baseline to 24 hours after segmental LPS challenge with endotoxin in the lung between CSL324 and placebo | Baseline to 24 hours after segmental LPS challenge with endotoxin in the lung
  Biomarkers are (neutrophil elastase [NE], alpha [α] 1 antitrypsin [AAT) complex, and myeloperoxidase [MPO]) in BALF
Percent reduction in the mean change in total protein in BALF from Baseline to 24 hours after segmental LPS challenge with endotoxin in the lung between CSL324 and placebo | Baseline to 24 hours after segmental LPS challenge with endotoxin in the lung
Percent reduction in the mean change in concentrations of von Willebrand factor (vWF) in BALF from Baseline to 24 hours after segmental LPS challenge with endotoxin in the lung between CSL324 and placebo | Baseline to 24 hours after segmental LPS challenge with endotoxin in the lung
Percent reduction in the mean change in concentrations of surfactant protein D (SP D) in BALF from Baseline to 24 hours after segmental LPS challenge with endotoxin in the lung between CSL324 and placebo | Baseline to 24 hours after segmental LPS challenge with endotoxin in the lung
Percent reduction in the mean change in concentrations of sRAGE in BALF from Baseline to 24 hours after segmental LPS challenge with endotoxin in the lung between CSL324 and placebo | Baseline to 24 hours after segmental LPS challenge with endotoxin in the lung
Percent reduction in the mean change in concentrations of G CSF in BALF from Baseline to 24 hours after segmental LPS challenge with endotoxin in the lung between CSL324 and placebo | Baseline to 24 hours after segmental LPS challenge with endotoxin in the lung
Percent reduction in the mean change in concentrations of VEGF A in BALF from Baseline to 24 hours after segmental LPS challenge with endotoxin in the lung between CSL324 and placebo | Baseline to 24 hours after segmental LPS challenge with endotoxin in the lung
Serum concentration of CSL324 | Up to 6 days after CSL324 administration
Number of subjects with antidrug antibodies (ADAs) to CSL324 in serum | Prior to and up to 6 days after CSL324 and placebo administration
Number and percentage of subjects with treatment-emergent adverse events (TEAEs) by treatment group | Up to 32 days after CSL324 and placebo administration
Maximum plasma concentration (Cmax) | Prior to and up to 6 days after CSL324 administration
Time to reach Cmax (Tmax) | Prior to and up to 6 days after CSL324 administration
Area under the plasma concentration-time curve from time 0 to 120 hours (AUC0-120h) | Time 0 to 120 hours after CSL324 administration
Area under the plasma concentration-time curve from time 0 to the last measurable concentration (AUC0-last) | Time 0 and up to 6 days after CSL324 administration

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (1):
- Fraunhofer Institute for Toxicology and Experimental Medicine, Hanover, Germany

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (ie FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.